CLINICAL TRIAL: NCT04530448
Title: Coronavirus Induced Acute Kidney Injury: Prevention Using Urine Alkalinization
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit enough subjects to complete the study. Only 3 subjects enrolled. However, those subjects did not complete the study as the PI terminated the study and data was not collected.
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005006707
Record Dates: First submitted 2020-08-20; First posted 2020-08-28 (Actual); Results first posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: COVID; Coronavirus; Coronavirus Infection; AKI; Acute Kidney Injury
Keywords: Acute Kidney Injury; AKI; COVID-19; Coronavirus; Sodium Bicarbonate
MeSH Terms: conditions — Coronavirus Infections; Acute Kidney Injury; COVID-19 | interventions — Sodium Bicarbonate; Standard of Care

STUDY DESIGN:
Intervention Model Description: Group 1 (control) will receive standard of care treatment for coronavirus according to institutional protocols.
  Group 2 (treatment) will receive sodium bicarbonate 225 mEq (225 mL of an 8.4% solution) intravenously over 1 hour.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of Care (Active Comparator): Standard of Care treatment
  Interventions: Other: Standard of Care
- Sodium Bicarbonate (Active Comparator): Sodium bicarbonate 225 mEq (225 mL of an 8.4% solution) intravenously over 1 hour. Sodium bicarbonate 8.4% solution should not exceed 900 ml (4 boluses) in 24 hours.
  Interventions: Drug: Sodium bicarbonate

INTERVENTIONS:
Drug: Sodium bicarbonate — Sodium bicarbonate 225 mEq (225 mL of an 8.4% solution) intravenously over 1 hour. Sodium bicarbonate 8.4% solution should not exceed 900 ml (4 boluses) in 24 hours.
  Arms: Sodium Bicarbonate
Other: Standard of Care — Standard of Care treatment
  Arms: Standard of Care

SUMMARY:
Our overarching goal is to improve the outcomes of critically ill COVID-19 patients with or at risk for development of acute kidney injury (AKI). The objective of this study is to determine the role of a protocol to manage urine alkalization using a simple medication that has been used for a very long time, is safe, and without significant side-effects. We aim to determine the feasibility and safety of a urine alkalinization protocol for the prevention of AKI in patients testing positive for COVID-19.

DETAILED DESCRIPTION:
Emerging evidence suggests that acute kidney injury (AKI) secondary to COVID-19 (COV-AKI) might result from direct infection of renal tubule epithelial cells (RTEC). A variety of epithelial cells express the ACE2 receptor which contains the receptor-binding domain (RBD) used by SARS-CoV-1 and SARS-CoV-2 to enter the cells. While direct infection of RTEC has not yet been proven data from multiple laboratories show virus in the kidney. It is this direct viral involvement of the RTEC that this proposal seeks to address.

One relatively simple approach would be to perturb the ability of the RBD to bind to its cellular (hACE2) receptor. Changes in pH may cause each amino acid residue, in the RBD, to assume a slightly different 'microscopic' conformation-dependent pKa value. Urine pH is normally 5.5- 6.5 (not too dissimilar to alveolar fluid-6.4-6.86) and can be easily and safely manipulated. In fact, urine alkalinization protocols have been used for decades to reduce renal toxicity from various compounds (especially chemotherapy) and are recommended by US and European toxicology societies. Here, the strategy will be deployed not for ion trapping but to inhibit the virus from infecting RTEC. Alkalinizing the urine using IV sodium-bicarbonate solution to pH of 7.5 or more can be easily and safely achieved.

While severe AKI does not appear to be a major part of the SARS-CoV-2 syndrome for most patients, when severe AKI does occur, mortality is very high and preventing early AKI may reduce AKI severity as the disease progresses.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 positive
* Admission to ICU or step-down unit
* Age ≥ 18 years old

Exclusion Criteria:

* Stage 3 AKI by KDIGO criteria
* CKD stage 4-5
* Contraindications to Na bicarbonate therapy (e.g. met. alkalosis, severe heart failure)
* Urine pH > 7.0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ankit Sakhuja, MD, Principal Investigator — West Virginia University
Locations (1):
- WVU Medicine Heart & Vascular Institute, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arentz M, Yim E, Klaff L, Lokhandwala S, Riedo FX, Chong M, Lee M. Characteristics and Outcomes of 21 Critically Ill Patients With COVID-19 in Washington State. JAMA. 2020 Apr 28;323(16):1612-1614. doi: 10.1001/jama.2020.4326. PMID 32191259
- [Background] Ali T, Khan I, Simpson W, Prescott G, Townend J, Smith W, Macleod A. Incidence and outcomes in acute kidney injury: a comprehensive population-based study. J Am Soc Nephrol. 2007 Apr;18(4):1292-8. doi: 10.1681/ASN.2006070756. Epub 2007 Feb 21. PMID 17314324
- [Background] Al-Jaghbeer M, Dealmeida D, Bilderback A, Ambrosino R, Kellum JA. Clinical Decision Support for In-Hospital AKI. J Am Soc Nephrol. 2018 Feb;29(2):654-660. doi: 10.1681/ASN.2017070765. Epub 2017 Nov 2. PMID 29097621
- [Background] Hoste EA, Bagshaw SM, Bellomo R, Cely CM, Colman R, Cruz DN, Edipidis K, Forni LG, Gomersall CD, Govil D, Honore PM, Joannes-Boyau O, Joannidis M, Korhonen AM, Lavrentieva A, Mehta RL, Palevsky P, Roessler E, Ronco C, Uchino S, Vazquez JA, Vidal Andrade E, Webb S, Kellum JA. Epidemiology of acute kidney injury in critically ill patients: the multinational AKI-EPI study. Intensive Care Med. 2015 Aug;41(8):1411-23. doi: 10.1007/s00134-015-3934-7. Epub 2015 Jul 11. PMID 26162677
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Wang HE, Muntner P, Chertow GM, Warnock DG. Acute kidney injury and mortality in hospitalized patients. Am J Nephrol. 2012;35(4):349-55. doi: 10.1159/000337487. Epub 2012 Apr 2. PMID 22473149
- [Background] Ponte B, Felipe C, Muriel A, Tenorio MT, Liano F. Long-term functional evolution after an acute kidney injury: a 10-year study. Nephrol Dial Transplant. 2008 Dec;23(12):3859-66. doi: 10.1093/ndt/gfn398. Epub 2008 Jul 15. PMID 18632586
- [Background] Collister D, Pannu N, Ye F, James M, Hemmelgarn B, Chui B, Manns B, Klarenbach S; Alberta Kidney Disease Network. Health Care Costs Associated with AKI. Clin J Am Soc Nephrol. 2017 Nov 7;12(11):1733-1743. doi: 10.2215/CJN.00950117. Epub 2017 Oct 19. PMID 29051143
- [Background] Sakhuja A, Kumar G, Gupta S, Mittal T, Taneja A, Nanchal RS. Acute Kidney Injury Requiring Dialysis in Severe Sepsis. Am J Respir Crit Care Med. 2015 Oct 15;192(8):951-7. doi: 10.1164/rccm.201502-0329OC. PMID 26120892
- [Background] Kellum JA, Prowle JR. Paradigms of acute kidney injury in the intensive care setting. Nat Rev Nephrol. 2018 Apr;14(4):217-230. doi: 10.1038/nrneph.2017.184. Epub 2018 Jan 22. PMID 29355173
- [Background] Tai W, He L, Zhang X, Pu J, Voronin D, Jiang S, Zhou Y, Du L. Characterization of the receptor-binding domain (RBD) of 2019 novel coronavirus: implication for development of RBD protein as a viral attachment inhibitor and vaccine. Cell Mol Immunol. 2020 Jun;17(6):613-620. doi: 10.1038/s41423-020-0400-4. Epub 2020 Mar 19. PMID 32203189
- [Background] Ren X, Glende J, Al-Falah M, de Vries V, Schwegmann-Wessels C, Qu X, Tan L, Tschernig T, Deng H, Naim HY, Herrler G. Analysis of ACE2 in polarized epithelial cells: surface expression and function as receptor for severe acute respiratory syndrome-associated coronavirus. J Gen Virol. 2006 Jun;87(Pt 6):1691-1695. doi: 10.1099/vir.0.81749-0. PMID 16690935
- [Background] Su H, Yang M, Wan C, Yi LX, Tang F, Zhu HY, Yi F, Yang HC, Fogo AB, Nie X, Zhang C. Renal histopathological analysis of 26 postmortem findings of patients with COVID-19 in China. Kidney Int. 2020 Jul;98(1):219-227. doi: 10.1016/j.kint.2020.04.003. Epub 2020 Apr 9. PMID 32327202
- [Background] Imai Y, Kuba K, Rao S, Huan Y, Guo F, Guan B, Yang P, Sarao R, Wada T, Leong-Poi H, Crackower MA, Fukamizu A, Hui CC, Hein L, Uhlig S, Slutsky AS, Jiang C, Penninger JM. Angiotensin-converting enzyme 2 protects from severe acute lung failure. Nature. 2005 Jul 7;436(7047):112-6. doi: 10.1038/nature03712. PMID 16001071
- [Background] Srivastava J, Barber DL, Jacobson MP. Intracellular pH sensors: design principles and functional significance. Physiology (Bethesda). 2007 Feb;22:30-9. doi: 10.1152/physiol.00035.2006. PMID 17289928
- [Background] RAMACHANDRAN GN, RAMAKRISHNAN C, SASISEKHARAN V. Stereochemistry of polypeptide chain configurations. J Mol Biol. 1963 Jul;7:95-9. doi: 10.1016/s0022-2836(63)80023-6. No abstract available. PMID 13990617
- [Background] Wan Y, Shang J, Graham R, Baric RS, Li F. Receptor Recognition by the Novel Coronavirus from Wuhan: an Analysis Based on Decade-Long Structural Studies of SARS Coronavirus. J Virol. 2020 Mar 17;94(7):e00127-20. doi: 10.1128/JVI.00127-20. Print 2020 Mar 17. PMID 31996437
- [Background] Choudhury D, Tanner MG, McAughtrie S, Yu F, Mills B, Choudhary TR, Seth S, Craven TH, Stone JM, Mati IK, Campbell CJ, Bradley M, Williams CK, Dhaliwal K, Birks TA, Thomson RR. Endoscopic sensing of alveolar pH. Biomed Opt Express. 2016 Dec 13;8(1):243-259. doi: 10.1364/BOE.8.000243. eCollection 2017 Jan 1. PMID 28101415
- [Background] Proudfoot AT, Krenzelok EP, Vale JA. Position Paper on urine alkalinization. J Toxicol Clin Toxicol. 2004;42(1):1-26. doi: 10.1081/clt-120028740. PMID 15083932
- [Background] Kashani K, Al-Khafaji A, Ardiles T, Artigas A, Bagshaw SM, Bell M, Bihorac A, Birkhahn R, Cely CM, Chawla LS, Davison DL, Feldkamp T, Forni LG, Gong MN, Gunnerson KJ, Haase M, Hackett J, Honore PM, Hoste EA, Joannes-Boyau O, Joannidis M, Kim P, Koyner JL, Laskowitz DT, Lissauer ME, Marx G, McCullough PA, Mullaney S, Ostermann M, Rimmele T, Shapiro NI, Shaw AD, Shi J, Sprague AM, Vincent JL, Vinsonneau C, Wagner L, Walker MG, Wilkerson RG, Zacharowski K, Kellum JA. Discovery and validation of cell cycle arrest biomarkers in human acute kidney injury. Crit Care. 2013 Feb 6;17(1):R25. doi: 10.1186/cc12503. PMID 23388612
- [Background] Emlet DR, Pastor-Soler N, Marciszyn A, Wen X, Gomez H, Humphries WH 4th, Morrisroe S, Volpe JK, Kellum JA. Insulin-like growth factor binding protein 7 and tissue inhibitor of metalloproteinases-2: differential expression and secretion in human kidney tubule cells. Am J Physiol Renal Physiol. 2017 Feb 1;312(2):F284-F296. doi: 10.1152/ajprenal.00271.2016. Epub 2016 Dec 21. PMID 28003188
- [Background] Singbartl K, Formeck CL, Kellum JA. Kidney-Immune System Crosstalk in AKI. Semin Nephrol. 2019 Jan;39(1):96-106. doi: 10.1016/j.semnephrol.2018.10.007. PMID 30606411

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Unable to recruit enough subjects to complete the study. Only 3 subjects enrolled. However, those subjects did not complete the study as the PI terminated the study and data was not collected.
Period: Overall Study
Arm/Group | Standard of Care | Sodium Bicarbonate
Started | 3 | 0
Completed | 0 | 0
Not Completed | 3 | 0
Not completed — Physician Decision | 3 | 0

BASELINE CHARACTERISTICS:
Population: Unable to recruit enough subjects to complete the study. Only 3 subjects enrolled. However, those subjects did not complete the study as the PI terminated the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Sodium Bicarbonate | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Continuous [Median (Full Range); unit: years] | 55 [52 to 61] |  | 55 [52 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 0 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: pH
Description: Primary feasibility outcome will be the proportion of patients treated who achieve >50% of urine measurements pH ≥= 7.2 over the duration of treatment.
Time Frame: 10 days
Population: Unable to recruit enough subjects to complete the study. Only 3 subjects enrolled. However, those subjects did not complete the study as the PI terminated the study and data was not collected.
Arm/Group | Standard of Care | Sodium Bicarbonate
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Number of Days Alive Free of Stage 2-3 AKI
Description: Primary efficacy outcome will be the number of days alive and free of stage 2-3 AKI (up to 28) in each group.
Time Frame: 28 days post-treatment
Population: as for outcome 1
Arm/Group | Standard of Care | Sodium Bicarbonate
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Stage 2-3 AKI
Description: proportion of patients developing stage 2-3 AKI (or stage 3 if already at stage 2 at enrollment).
Time Frame: 28 days
Population: as for outcome 1
Arm/Group | Standard of Care | Sodium Bicarbonate
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Vent-Free
Description: Ventilator-free days to 28 days
Time Frame: 28 days
Population: as for outcome 1
Arm/Group | Standard of Care | Sodium Bicarbonate
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Hospital-Free
Description: Hospital-free days to 60 days
Time Frame: 60 days post-index hospitalization
Population: as for outcome 1
Arm/Group | Standard of Care | Sodium Bicarbonate
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 months
Description: Unable to recruit enough subjects to complete the study. Only 3 subjects enrolled in the Standard of Care Arm of the study. However, those subjects did not complete the study as the PI terminated the study.
Arm/Group | Standard of Care | Sodium Bicarbonate
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT04530448/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/48/NCT04530448/ICF_001.pdf